CLINICAL TRIAL: NCT06855043
Title: Pilot Randomized Controlled Trial of Late Surfactant Therapy With Budesonide for Prevention of Bronchopulmonary Dysplasia
Brief Title: Little Lungs Study
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Meriter Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1479; A536757 (Other: UW Madison); SMPH\PEDIATRICS\NEONATO (Other: UW Madison); Protocol Version 10/09/25 (Other: UW Madison)
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Invasive Mechanical Ventilation; Severe Respiratory Distress Syndrome
Keywords: premature birth
MeSH Terms: conditions — Respiratory Distress Syndrome; Premature Birth | interventions — calfactant; Budesonide

STUDY DESIGN:
Intervention Model Description: This is a phase I/II pilot randomized controlled clinical trial to obtain preliminary data on safety and clinical response of multiple doses of late surfactant treatment with budesonide
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Premature babies: Study Intervention (Experimental): Preterm infants born at gestational age less than 29 0/7 weeks requiring mechanical ventilation at 7-14 days of life (targeting N=12 participants completing study to 7 days post-intervention)
  Interventions: Drug: Calfactant; Drug: Budesonide
- Premature babies: Standard of Care (No Intervention): Preterm infants born at gestational age less than 29 0/7 weeks requiring mechanical ventilation at 7-14 days of life (targeting N=12 participants completing study to 10 days post-randomization)

INTERVENTIONS:
Drug: Calfactant — Participants will receive 2 daily doses of Calfactant (3 ml/kg) intratracheal administration
  Arms: Premature babies: Study Intervention
Drug: Budesonide — Participants will receive 2 daily doses of Budesonide (0.25mg/kg) intratracheal administration.
  Arms: Premature babies: Study Intervention

SUMMARY:
This clinical trial is being done to evaluate the safety and clinical response of late surfactant treatment with budesonide in extremely preterm infants requiring mechanical ventilation at 7-14 days of age.

DETAILED DESCRIPTION:
Primary Objective

• To evaluate safety of late surfactant therapy with budesonide in extremely preterm infants.

Secondary Objectives

* To evaluate the oxygenation response to late surfactant therapy with budesonide in extremely preterm infants at 48 hours and 7 days after completion of the study intervention
* To evaluate respiratory outcomes following administration of late surfactant therapy with budesonide

ELIGIBILITY:
Neonate Inclusion Criteria:

* Gestational age 22 0/7 to 28 6/7 weeks at birth
* Age 7-14 days
* Need invasive mechanical ventilatory support and a Fraction of Inspired Oxygen (FiO2) greater than or equal to 0.3

Birthing Parent Inclusion Criteria:

* Have a baby who meets neonate eligibility criteria and enrolls in the study.

Neonate Exclusion Criteria:

* Major congenital anomalies including congenital lung malformations and congenital diaphragmatic hernia and/or genetic disorders
* Alternative, acute clinical etiology of respiratory deterioration or increased ventilatory requirements (e.g., sepsis, pneumonia, etc.)
* History of pulmonary hemorrhage
* Antibiotic use within 48 hours
* Indomethacin or Ibuprofen use within 72 hours
* Prior treatment with corticosteroids for prevention of lung disease
* Not expected to survive for greater than 7 days at enrollment
* Determined to be unstable by the clinical team
* Enrolled in a conflicting clinical trial
* Have a birth parent aged less than 18 years
* Parent/guardian is unable to provide parental permission in English or Spanish

Ages: 7 Days to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2026-09 (Estimated); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of acute clinical deterioration up to 60 minutes after study intervention | up to 60 minutes after study intervention (intervention received within 14 days of life (DOL))
  Presence or absence of acute clinical deterioration - defined as desaturation less than 80 percent and/or bradycardia less than 100 beats per minute (bpm) - during the study intervention and up to 60 minutes after study intervention.
Presence or absence of severe acute clinical deterioration up to 60 minutes after study intervention | up to 60 minutes after study intervention (intervention received within 14 DOL)
  Presence or absence of severe acute clinical deterioration - defined as desaturation less than 60 percent and/or bradycardia less than 80 bpm - during the study intervention and up to 60 minutes after study intervention.
Occurrence of pneumothorax needing evacuation up to 48 hours after completion of study intervention | baseline to 48 hours after completion of study intervention (intervention received within 14 DOL)
  A yes or no question of whether there was pneumothorax (air in the pleural cavity) detected via chest x-ray, needing evacuation from baseline to 48 hours after completion of study intervention
Occurrence of pulmonary hemorrhages up to 48 hours after completion of study intervention | baseline to 48 hours after completion of study intervention (intervention received within 14 DOL)
  A yes or no question of whether pulmonary hemorrhage (bleeding in lungs) was observed in the endotracheal tube from baseline to 48 hours after completion of study intervention.

SECONDARY OUTCOMES:
Change in Respiratory Severity Score (RSS) | Baseline to 7 days post-intervention (intervention received within 14 DOL)
  RSS is the mean airway pressure multiplied by the fraction of inspired oxygen, a change toward higher scores indicates more severe respiratory symptoms.
Death or Grade 3 Bronchopulmonary Dysplasia (BPD) by 36 0/7 weeks Post-Menstrual Age (PMA) | up to 36 0/7 weeks PMA
Days of mechanical ventilation by 36 0/7 weeks PMA | up to 36 0/7 weeks PMA
  Days of mechanical ventilation by 36 0/7 weeks PMA (If an infant died before 36 0/7 weeks, time from death to 36 0/7 weeks PMA will be considered as mechanical ventilation days)

CONTACTS AND LOCATIONS:
Overall Officials: Dinushan Kaluarachchi, MBBS, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - Meriter Hospital, Madison, Wisconsin
  - American Family Children's Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF